CLINICAL TRIAL: NCT04878510
Title: Non-invasive Ventilation and Dexmedetomidine in Critically Ill Adults: a Vanguard Pragmatic Randomized Controlled Trial (inDEX Trial)
Brief Title: Non-invasive Ventilation and Dex in Critically Ill Adults
Acronym: inDEX
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: St. Joseph's Healthcare Hamilton (Other)
Responsible Party: Principal Investigator, Kimberley Lewis, Clinical Scholar; Principal Investigator, St. Joseph's Healthcare Hamilton
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 13205
Record Dates: First submitted 2021-04-25; First posted 2021-05-07 (Actual); Last update posted 2024-10-28 (Actual); Status verified 2024-10

CONDITIONS: Respiratory Insufficiency
Keywords: Non-Invasive Ventilation; Sedation; Randomized Control Trial; Acute Respiratory Failure
MeSH Terms: conditions — Respiratory Insufficiency | interventions — Dexmedetomidine

STUDY DESIGN:
Intervention Model Description: The inDEX trial is a pragmatic, international, multi-centered, stratified, randomized, parallel-group, double-blind, placebo-controlled vanguard trial.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: To minimize performance and ascertainment biases, and maintain blinding of patients, investigators, clinical staff, and research coordinators; a Research Pharmacist, who is not involved in assessment of patient outcomes or patient care, will prepare infusion bags
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dexmedetomidine Intervention (Experimental): Patients randomized to the experimental arm will receive dexmedetomidine. At initiation, a bolus will NOT be administered. In keeping with Health Canada. Guidelines, the infusion will start at a mid-range dose of 0.6mcg/kg/h with titration either up or down by 0.1mcg/kg/h every 20-30 minutes to a maximum rate of 1.2mcg/kg/h to maintain light sedation (Richmond Agitation-Sedation Scale [RASS] = -2 to +1 or Riker Sedation-Agitation Scale [SAS] 3-4).
  Interventions: Drug: Dexmedetomidine
- Control Intervention (Placebo Comparator): Those in the control group will receive a placebo that is identical in colour and packaging and at equal volume to the intervention group. Each bag of placebo contains 50mL of 0.9% sodium chloride and labeled as per Health Canada guidance for labelling pharmaceutical drugs for use in humans.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Dexmedetomidine — Dexmedetomidine is an α2-adrenergic agonist sedative commonly used in invasive mechanical ventilation that promotes patient wakefulness, has no effect on respiratory drive, has important analgesic properties, and when compared to γ-aminobutyric acid receptor agonists like benzodiazepines, reduces delirium.
  Other Names: Precedex
  Arms: Dexmedetomidine Intervention
Other: Placebo — Normal saline placebo will be given as continuous infusion.
  Arms: Control Intervention

SUMMARY:
Non-Invasive ventilation (NIV) is a life saving intervention for patients with acute respiratory failure (ARF). Some patients are not able to tolerate the NIV intervention and ultimately fail, requiring the use of invasive mechanical ventilation (IMV) and intubation. Sedation may improve a patient's NIV tolerance. However, this practice has not been adopted by intensivists as the risk of over-sedation resulting in respiratory depression, inability to protect the airway, and inadvertent need for intubation are all large deterrents of sedative use in NIV.

The Non-invasive Ventilation and Dexmedetomidine in Critically Ill Adults: a Vanguard Pragmatic Randomized Controlled Trial (inDEX) is looking to evaluate the effectiveness of dexmedetomidine compared to placebo in reducing non-invasive ventilation failures in patients admitted to the hospital with acute respiratory failure. The results from this pilot trial, will subsequently inform a large, pragmatic, powered trial to definitively address the question.

DETAILED DESCRIPTION:
1. BACKGROUND:

   Non-invasive ventilation (NIV) is a life-saving intervention for patients with acute respiratory failure (ARF). Patients may find NIV intolerable and ultimately fail NIV requiring intubation and invasive mechanical ventilation (IMV). Sedation may improve a patient's NIV tolerance. However, this practice has not been adopted by intensivists as the risk of over-sedation resulting in respiratory depression, inability to protect the airway, and inadvertent need for intubation are all large deterrents of sedative use in NIV. Current guidelines lack recommendations on which sedative, if any at all, should be used during NIV due to the paucity of reliable data. Dexmedetomidine (dex) is a relatively new sedative. It promotes patient wakefulness, has no effect on respiratory drive, has important analgesic properties, and when compared to γ-aminobutyric acid receptor agonists like benzodiazepines, reduces delirium. Dex has been recommended to use over benzodiazepines for sedation during IMV in critically ill adults, particularly if delirium is precluding weaning.
2. HYPOTHESIS:

   We hypothesize that dexmedetomidine, when compared to placebo, reduces NIV failure in hospitalized adults with acute respiratory failure and agitation or NIV intolerance.
3. OBJECTIVES:

   To evaluate the feasibility of assessing if dexmedetomidine compared to placebo results in a reduction of non-invasive ventilation failure in patients admitted to the hospital with acute respiratory failure. This will subsequently inform a large, pragmatic, powered trial to definitively address the question.
4. METHODS

4.1 Study design: The inDEX trial is a pragmatic, international, multi-centered, stratified, randomized, parallel-group, double-blind, placebo-controlled vanguard trial. Patients, investigators, healthcare team, data collectors, outcome assessors, and the statistician will be blinded to trial arms.

4.2 Allocation and randomization: Local Research Coordinators (RC) will randomize eligible patients in a fixed 1:1 allocation using undisclosed variable block sizes of four, six, or eight. The randomization will be achieved using a random number sequence prepared by an independent statistician. The independent statistician will have access to the random number sequence and it will be provided to the research pharmacist. Upon request by the local research coordinator, the research pharmacist will provide the care team with either placebo or dexmedetomidine, according to the randomization schedule. 4.3 Blinding: Both dexmedetomidine and normal saline placebo will be given as continuous infusion. To minimize performance and ascertainment biases, and maintain blinding of patients, investigators, clinical staff, and RCs; a Research Pharmacist, who is not involved in assessment of patient outcomes or patient care, will prepare infusion bags. Titration of the infusion rate for both arms will follow an identical volume-based titration algorithm. Despite optimal blinding efforts, it is possible that the care team may be able to determine who is receiving dexmedetomidine based on improvement in NIV tolerance and/or the decrease in heart rate and blood pressure. However, the cointerventions may also improve tolerance, and can certainly cause a reduction in heart rate and blood pressure.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years
2. Patient receiving any NIV modality for acute respiratory failure of any etiology
3. Admitted to ICU, PACU, step-down unit (surgical or medical), or emergency department
4. Presence of one or more of the following after optimized NIV treatment

   1. Agitation (Defined as a Richmond Agitation and Sedation Scale [RASS] score of ≥+2 or a Riker Sedation-Agitation Scale [SAS] score of ≥5)
   2. Patient expresses intolerance or requests removal of NIV secondary to self-reported discomfort, anxiety, or claustrophobia
   3. Other reason that the physician feels the patient is intolerant of NIV or agitated, not captured above (all reasons will be recorded)

Exclusion Criteria:

1. Absence of a functioning pacemaker with one of the following: a-Persistent bradycardia defined as a heart rate (HR) ≤50bpm; b-Second or third-degree heart block; or c- Tachybrady syndrome
2. Persistent hypotension, defined as a mean arterial pressure (MAP) ≤60mmHg despite volume resuscitation and vasopressors
3. Acute hepatic failure
4. Known allergy to dexmedetomidine
5. Pregnancy
6. Acute withdrawal from drugs or alcohol
7. Patients with post-extubation respiratory failure
8. Imminent need for endotracheal intubation
9. Death is deemed imminent and inevitable
10. Patient's goals of care do not include intubation and IMV
11. Patients already on dexmedetomidine at time of enrollment
12. Previously enrolled in the inDEX trial
13. Treating physician refuses enrollment (reasons for refusal will be captured)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2022-03-07 (Actual); Primary Completion 2024-04-21 (Actual); Study Completion 2024-04-21 (Actual)

PRIMARY OUTCOMES:
Recruitment Rate | At the completion of the trial (approximately 1 year).
  The rate in which patients are enrolled, by calculating the mean number of recruited patients compared to the number of patients screened.
Protocol Adherence; Proportion of patients assigned to the experimental arm that received the intervention and those assigned to the control arm that did not receive the intervention. | At the completion of the trial (approximately 1 year).
  Adherence will be calculated as the proportion of patients assigned to the experimental arm that received the intervention and those assigned to the control arm that did not receive the intervention.
Consent Rate | At the completion of the trial (approximately 1 year).
  The consent rate will be calculated as the overall proportion of substitute decision makers or patients who consented to be enrolled out of those approached.

SECONDARY OUTCOMES:
Acute care unit outcomes; Non-invasive ventilation (NIV) failure | 28 days post-randomization.
  Number of participants with NIV failure defined as the patients undergoing invasive mechanical ventilation within 28-post randomization.
Acute care unit outcomes; Acute Care Unite Length of Stay | 60 days post-randomization.
  Acute Care Unite Length of Stay is defined as the number of days the patient is admitted to an Acute Care Unit while admitted to the hospital.
Acute care unit outcomes; Duration of invasive mechanical ventilation | 60 days post-randomization.
  Duration of invasive mechanical ventilation during hospital stay is defined as the number of days the patient received invasive mechanical ventilation at 60 days post-randomization.
Acute care unit outcomes; Ventilation free Days | 28 days post-randomization.
  Ventilation free days is defined as the number of days the patient did not receive and ventilation during hospital stay truncated at 28 days (either invasive mechanical ventilation or NIV).
Process Outcomes; Number of patient-initiated device removal episodes. | 4 days post-randomization.
  Number of patient-initiated device removal episodes will be defined as the number of times a patient attempts to remove their device while receiving NIV.
Process Outcomes; Richmond-Agitation Sedation Scale (RASS) measurements | 4 days post-randomization.
  The proportion of RASS measurements in target range while on the trial drugs while receiving NIV.
Process Outcomes; The mean NIV tolerance score. | 4 days post-randomization.
  The mean NIV tolerance score will be defined as the proportion of tolerance scores that indicate that the patient is comfortable and relaxed while receiving NIV.
Process Outcomes; Days spent with delirium | 28 days post-randomization.
  Days spent with delirium will be defined as the number of days that the patient experienced delirium during and after receiving NIV while admitted to the hospital.
Process Outcomes; Cointerventions | 4 days post-randomization.
  The use and dose of any cointerventions (i.e. benzodiazepines, opioids, and antipsychotics) during NIV treatment.
Hospital Outcomes; Hospital length of stay | 60 days post-randomization.
  Hospital Length of stay is defined at the total number of days the patient spent in the hospital.
Hospital Outcomes; Mortality | 60 days post-randomization.
  Mortality is defined at the number of deaths that occur between randomization and 60-Day post-randomization.
Adverse Events: Bradycardia | 60 Days post-randomization
  Adverse events will be defined as; bradycardia (heart rate <60 bpm).
Adverse Events: Severe bradycardia | 60 Days post-randomization
  Adverse events will be defined as; severe bradycardia (heart rate <50 bpm).
Adverse Events: Clinically significant bradycardia | 60 Days post-randomization
  Adverse events will be defined as; clinically significant bradycardia (bradycardia requiring inotropes, vasopressors, external pacing, temporary pacemaker, or discontinuation of the trial medication).
Adverse Events: hypotension | 60 Days post-randomization
  Adverse events will be defined as; hypotension (mean arterial pressure < 60mmHg, or >20mmHg below admission baseline).
Adverse Events: clinically significant hypotension | 60 Days post-randomization
  Adverse events will be defined as; clinically significant hypotension (hypotension requiring vasopressors, fluid administration, or discontinuation of the trial medication).
Adverse Events: hypertension | 60 Days post-randomization
  Adverse events will be defined as; hypertension (a systolic blood pressure >180mmHg or a diastolic blood pressure >110mmHg).
Adverse Events: Cardiac Arrest | 60 Days post-randomization
  Adverse events will be defined as; cardiac arrest.
Functional Outcomes; quality of life | 60 Days post-randomization
  Functional Outcomes will be defined as; quality of life outcomes will be collected using the EQ-5D-5L questionnaire at pre-hospital, baseline, 28-Days and 60-Days post-randomization.
Functional Outcomes; clinical frailty | 60 Days post-randomization
  Functional Outcomes will be defined as the "clinical frailty score" will be collected at pre-hospital, baseline, 28-Days and 60-Days post-randomization.

CONTACTS AND LOCATIONS:
Overall Officials: Kimberley Lewis, MD, Principal Investigator — Research Institute of St Joseph's Healthcare Hamilton
Locations (3):
- Monash Medical Centre - Monash Health, Melbourne, Australia
- St. Joseph's Healthcare Hamilton, Hamilton, Ontario, Canada
- King Abdulaziz Medical City - Riyadh, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No